CLINICAL TRIAL: NCT00165646
Title: A Double-Blind, Placebo-Controlled, Comparative Study on the Efficacy and Safety of E3810 in Patients With Non-erosive Gastroesophageal Reflux Disease
Brief Title: A Comparative Study on the Efficacy and Safety of E3810 in Patients With Non-erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Nobuyuki Sugisaki, Eisai Co., Ltd.
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-J081-461
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2010-08

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease
Keywords: non-erosive gastroesophageal reflux disease; NERD; proton pump inhibitor; rabeprazole
MeSH Terms: interventions — Rabeprazole

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: E3810
- 2 (Experimental)
  Interventions: Drug: E3810
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E3810 — E3810 5mg: once daily orally for 4 weeks
  Arms: 1
Drug: E3810 — E3810 10mg: once daily orally for 4 weeks
  Arms: 2
Drug: Placebo — Placebo: once daily orally for 4 weeks
  Arms: 3

SUMMARY:
To investigate the efficacy and safety of a 4-week treatment of 5 mg/day or 10 mg/day of E3810 (Pariet (Rabeprazole Sodium)) in patients with non-erosive gastroesophageal reflux disease in a multicenter, randomized, double-blind, comparative study.

ELIGIBILITY:
Inclusion Criteria:

The patients to be included will be outpatients who meet all of the following criteria. No specific gender is asked.

<For the observation period>

1. Patients who have "heartburn" 2 days a week or more for consecutive weeks during 3 weeks prior to pre-observation screening. If a day of screening and a day of starting observation (date of registration) are different, heartburn must continuously be present during the in-between period.
2. Patients who meet both 1) and 2) below; 1) The symptom is a burning sensation arising from the stomach or the lower chest.

2) The symptom tends to appear frequently or is aggravated after eating, when bending a body forward, and/or when pressing on the abdomen.

(3) Patients categorized in "grade M" (discoloring type: minimal change) according to the Los Angeles System (2nd Modification) for Classification of Reflux Esophagitis.

(4) Patients who are 20 years old or older at the time of obtaining consent. (5) Patients who are informed of the objective and details of the study and give written consent for study entry.

<For the treatment period>

1. Patients who have "heartburn" on 2 days a week or more in 7 days immediately before the treatment period (during the observation period).
2. Patients with "heartburn diary" that is completely filled out for 7 days until the treatment period (during the observation period). If the observation period is 8 days or longer, those with heartburn diary of which entries are fulfilled 80% or more during the observation period.
3. Patients with 80% or better drug compliance for antacids during the observation period.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study.

1. Patients who cannot keep adequate entries of heartburn diary by themselves.
2. Patients who strongly complain "feeling of heavy stomach" and/or "abdominal bloating."
3. Patients who have a complication or history of psychiatric or psychosomatic disease (e.g., manic-depressive psychosis, obsessive-compulsive neurosis, or others) or those who are on an antidepressant or anti-anxiety agent (accepted if only for a hypnotic treatment).
4. Patients who have undergone Helicobacter pylori eradication therapy, and less than 6 months have elapsed from the end of H. pylori eradication therapy to the beginning of the observation period. : The same day 6 months earlier, and the day at the end of 6 months earlier if it is at the end of month.
5. Patients with open gastric or duodenal ulcer.
6. Patients with acute gastritis.
7. Patients with a history of any surgical intervention that affect peptic secretion (e.g., upper gastrointestinal tract resection and/or vagotomy).
8. Patients with Barrett's esophagus, esophageal stenosis, or pyloric stenosis.
9. Patients with scleroderma.
10. Patients with a history or complication of angina pectoris.
11. Patients who work at night (working for a night-shift).
12. Patients who received proton pump inhibitors (PPIs) within 3 weeks prior to pre-observation screening
13. Patients who need NSAIDs (except topical preparations), steroids (except topical preparations), and/or aspirin treatment every day
14. Patients receiving dialysis therapy
15. Patients with a serious complication such as cardiovascular disease (e.g., myocardial infarction), hematological disorder (e.g., aplastic anemia), renal disease (e.g., acute or chronic renal failure), hepatic disease (e.g., cirrhosis), or malignant tumor.
16. Patients with known hypersensitivity to antacids or PPIs.
17. Patients who are pregnant or those with childbearing potential, or those who wish to become pregnant or are lactating during the study period.
18. Patients receiving another investigational drug or those who received another investigational drug within 6 months prior to pre-observation screening : Registration is allowed on the same day of 6 months earlier, and the day at the end of 6 months earlier if it is at the end of month.
19. Patients who are judged to be ineligible for the study entry by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2004-09; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sugisaki, Study Director — Eisai Co., Ltd - Development Clinical Research Department. Clinical Research Center
Locations (23):
- Japan (23):
  - Aichi-Gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Chikushino-shi, Fukuoka
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Maebashi, Gunma
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido-Prefecture
  - Kochi, Kochi
  - Kyoto, Kyoto
  - Sandai, Miyagi
  - Sendai, Miyagi
  - Moriguchi, Osaka
  - Osaka, Osaka
  - Saga, Saga-ken
  - Kawaguchi, Saitama
  - Izumo, Shimane
  - Matsue, Shimane
  - Hamamatsu, Shizuoka
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Sanyōonoda, Yamaguchi
  - Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 35 centers in Japan during the period of Sep-2004 to Oct-2005.
Pre-assignment Details: Antacid was administered 1-2 weeks for observational period (non-blind). Patients showing the resistance to antacid were transferred to treatment period (randomized double-blind) of placebo, E3810 5 or 10 mg/day for four weeks.
Groups:
- Placebo: once daily orally for 4 weeks
- E3810 5 mg: E3810 (Pariet (Rabeprazole Sodium)) 5 mg once daily orally for 4 weeks
- E3810 10 mg: E3810 (Pariet (Rabeprazole Sodium))10 mg once daily orally for 4 weeks
Period: Overall Study
Arm/Group | Placebo | E3810 5 mg | E3810 10 mg
Started | 93 | 93 | 102
Completed | 88 | 88 | 98
Not Completed | 5 | 5 | 4
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Physician Decision | 2 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | E3810 5 mg | E3810 10 mg | Total
Number analyzed (Participants) | 91 | 93 | 101 | 285
Age Continuous [Mean (Standard Deviation); unit: years] — Full Analysis Set Population
  years | 49.7 (17.0) | 46.3 (15.3) | 46.8 (15.7) | 47.6 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 55 | 51 | 157
  Male | 40 | 38 | 50 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Asian | 91 | 93 | 101 | 285
Region of Enrollment [Number; unit: participants]
  Japan | 91 | 93 | 101 | 285

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Relief of Heartburn at Final Evaluation
Description: "Heartburn diary" will be given to each subject and ask him/her to keep the diary every day throughout the study period. The subject will be requested to record the occurrence of heartburn during the daytime and the nighttime in the diary. Primary End Point is the rate of complete disappearance of heartburn. The rate of heartburn do not occur in the past week will be calculated based on the diary. Participants were evaluated at week 4 about episodes of heartburn in the last 7 days
Time Frame: 4 weeks
Population: The major endpoint of this study was between-group comparison of the complete relief of heartburn (at the completion of the treatment period) in the full analysis set (FAS).
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | E3810 5 mg | E3810 10 mg
Number analyzed (Participants) | 91 | 93 | 101
Percentage of participants | 20.9 | 34.4 | 43.6

ADVERSE EVENTS:
Arm/Group | Placebo | E3810 5 mg | E3810 10 mg
Serious Adverse Events (participants affected / at risk) | 0/91 | 1/93 | 0/102
Other Adverse Events (participants affected / at risk) | 32/91 | 32/93 | 37/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | E3810 5 mg (N=93) | E3810 10 mg (N=102)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 | 1 | 0 — These AEs occurred 23days after the end of administration.
Reflux oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 — These AEs occurred 23days after the end of administration.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | E3810 5 mg (N=93) | E3810 10 mg (N=102)
Nasopharyngitis (Infections and infestations) | 9 (9) | 6 (7) | 4 (4)
Cystitis (Infections and infestations) | 0 | 0 (0) | 2 (3)
Bronchitis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Acute tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia oral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 1 (1)
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 2 (2) | 1 (1) | 3 (3)
Malaise (General disorders) | 2 (2) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No